CLINICAL TRIAL: NCT03922360
Title: Smartphone-based Financial Incentives
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Allison N Kurti, Research Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRMS 17-0604
Record Dates: First submitted 2019-04-04; First posted 2019-04-19 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine Dependence; Financial Incentives; Pregnant Women; Smoking Cessation; mHealth; Smartphone
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Intervention Model Description: We are proposing a two condition, parallel groups, randomized controlled trial (RCT) of a mobile-phone-based financial incentives intervention targeting economically disadvantaged pregnant cigarette smokers. The experimental group will receive electronic vouchers contingent on the remote submission of breath carbon monoxide (CO) samples indicating smoking abstinence whereas the control group will receive best practices for promoting smoking cessation. The use of a best practices control group reflects a real-world comparison condition in that all women will receive the treatment that practitioners in the community are instructed to provide (i.e., the 5As plus quit-line referral) thereby enhancing the ecological validity of the study, while also minimizing between-subject variability in the extent of participants' exposure to these practices by implementing these treatment components ourselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Practices (Active Comparator)
  Interventions: Behavioral: Best Practices
- Best Practices + Financial Incentives (Experimental)
  Interventions: Behavioral: Smartphone-based Financial Incentives

INTERVENTIONS:
Behavioral: Smartphone-based Financial Incentives — Best Practices- The 2008 Clinical Practice Guidelines for smoking cessation recommends that pregnant smokers be provided with the 5As. Research staff will implement the 5As at three assessments that take place during pregnancy.
  Best Practices + Financial Incentive- Women assigned to this condition will receive the best practices treatment described above plus the remote incentives intervention.
  Beginning on the quit date and extending for one week, participants will be required to submit twice daily CO samples. All samples < 6 ppm will be considered negative and those > 6 ppm will be considered positive. Participants will earn incentives for breath tests indicating smoking abstinence, and incentive values will increase with each consecutive negative sample. Following the initial quit week, the schedule of monitoring will be reduced and incentives will be contingent on submitting a negative saliva cotinine test.
  Other Names: Contingency Management
  Arms: Best Practices + Financial Incentives
Behavioral: Best Practices — Best Practices- The 2008 Clinical Practice Guidelines for smoking cessation recommends that pregnant smokers be provided with the 5As. Research staff will implement the 5As at three assessments that take place during pregnancy.
  Arms: Best Practices

SUMMARY:
Cigarette smoking during pregnancy increases risk for catastrophic pregnancy complications, growth retardation, other adverse fetal and infant health problems, and later-in-life chronic conditions among exposed offspring. The most effective intervention for reducing smoking during pregnancy is financial incentives whereby participants earn incentives (e.g., gift cards, cash) contingent on objective evidence of smoking abstinence. However, financial incentives-based interventions are typically delivered in relatively intense protocols requiring frequent clinic visits, which limits the geographical range over which services can be delivered and potentially denies treatment to those residing in remote or otherwise difficult to reach settings.

The present study will examine the feasibility, efficacy, and cost-effectiveness of a smartphone-based financial incentives intervention whereby smoking monitoring and delivery of incentives are completed remotely using a mobile app (to be designed by DynamiCare Health, Inc.). Eligible participants who complete the informed consent process will be randomized to one of two conditions: an incentives condition wherein women will receive financial incentives contingent on the remote submission of breath and saliva specimens indicating abstinence from recent smoking (described below), or a best practices control condition in which women will receive usual care for smoking cessation that is provided at their obstetrical clinics, as well as three brief educational sessions and referral to the Vermont (or other state) pregnancy-specific quit line by our research staff.

For inclusion in the study, women must meet the following criteria: (a) > 18 years of age, (b) report being smokers at the time they learned of the current pregnancy, (c) report smoking in the 7 days prior to completing their phone eligibility screening, (c) < 25 weeks pregnant, (d) speak English, (e) own a smartphone (Android or iOS; 81.8% of pregnant women in wave 1 [2013-2014] of the Population Assessment of Tobacco and Health [PATH] reported owning a smartphone). Exclusion criteria include: (a) current or prior mental or medical condition that may interfere with study participation (assessed via self-report during phone eligibility screening), (b) smoke marijuana more than once each week and not willing to quit (marijuana smoking can inflate breath CO), (c) exposed to unavoidable occupational sources of CO (e.g., car mechanic), and (d) self-report currently being maintained on opioid maintenance therapy (e.g., methadone, buprenorphine).

Participants randomized to the incentives condition will select a quit date (either the first or second Monday following their enrollment), and will submit videos of themselves blowing into a breath CO monitor twice daily during week 1. They will receive incentives for every sample where expired breath CO is < 6 ppm. Beginning in week 2 and extending through week 6, participants will submit videos twice per week (Monday/Thursday) for which they will receive incentives for providing videos of themselves completing saliva cotinine tests indicating smoking abstinence. From week 7 until delivery, participants will submit videos once per week and will continue to receive incentives for saliva cotinine tests indicating no smoking. During the postpartum period, women will submit videos twice weekly for the first 4 weeks and once weekly from weeks 5-12. Women will receiving incentives for negative breath and saliva samples, and the value of incentives will increase with each consecutive sample indicating smoking abstinence. Participants will not receive incentives for missed samples or samples that indicate smoking, and the incentive schedule will be reset at its starting value. However two consecutive negative samples following a missed or positive sample will restore the incentive to its prior value.

Women in both conditions will complete seven formal assessments of their smoking status during their participation along with a treatment acceptability questionnaire and semi-structured interview on barriers and facilitators of treatment engagement.

We conducted a power analysis to estimate the number of participants required to detect treatment effects assuming late-pregnancy abstinence rates of approximately 40% vs. < 10% (incentives vs. best practices, respectively), and 24-week postpartum abstinence rates of approximately 20% vs. < 5%. The proposed sample size of 76 per treatment condition will result in at least 80% power to detect a difference between the two treatment conditions in abstinence rates of 40% vs. 10 % at late-pregnancy or 20% vs. 5% at 24-weeks postpartum assessments using a chi-square test and significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* report being smokers at the time they learned of the current pregnancy
* report smoking in the 7 days prior to completing their preliminary eligibility screening,
* < 25 weeks pregnant
* speak English
* own a smartphone

Exclusion Criteria:

* current or prior mental or medical condition that may interfere with study participation (assessed via self-report during formal intake assessment completed online or by phone using a medical and psychosocial history questionnaire)
* smoke marijuana more than once each week and not willing to quit (marijuana smoking can inflate breath CO)
* exposed to unavoidable occupational sources of CO (e.g., car mechanic)
* report currently receiving opioid maintenance therapy (e.g., methadone, buprenorphine).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Early Pregnancy Quit Rate | One month after participant's enrollment date
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
Late Pregnancy Quit Rate | 28 weeks gestation or later
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
4-week Postpartum Quit Rate | 4 weeks following the date that participants deliver their infant
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
8-week Postpartum Quit Rate | 8 weeks following the date that participants deliver their infant
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
12-week Postpartum Quit Rate | 12 weeks following the date that participants deliver their infant
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
24-week Postpartum Follow-up | 24 weeks following the date that participants deliver their infant
  Point prevalence smoking abstinence (defined as a cotinine-negative saliva test AND self-reported no smoking in the past seven days)
Longest Duration of Abstinence (LDA) | LDA will be measured from participant's date of enrollment in the study to 24-wks postpartum
  Consecutive days of no smoking using biochemical verification (cotinine-negative saliva at the formal assessments described above) plus self-report (cigarettes per day from enrollment to 24 wks postpartum reported during timeline follow-back conducted over the phone)
Mean birth weight | Participants sign a medical release for their infant's birth report prior to study enrollment. Fax requests for infant birth reports are submitted upon confirming actual delivery dates/locations with them or within 1 month of expected delivery dates
  Mean birth weight (in grams) as reported on delivery reports among infants born to mothers enrolled in the study
Gestational age at delivery | Participants sign a medical release for their infant's birth report prior to study enrollment. Fax requests for infant birth reports are submitted upon confirming actual delivery dates/locations with them or within 1 month of expected delivery dates
  Gestational age (in weeks) at delivery as reported on delivery reports among infants born to mothers enrolled in the study
NICU admissions | Participants sign a medical release for their infant's birth report prior to study enrollment. Fax requests for infant birth reports are submitted upon confirming actual delivery dates/locations with them or within 1 month of expected delivery dates
  Yes/no regarding whether infant was admitted to the NICU, and number of days in the NICU, as reported on delivery reports among infants born to mothers enrolled in the study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States